CLINICAL TRIAL: NCT01280526
Title: A Phase IB/II Study of Escalating Doses of Romidepsin (Istodax®) in Association With CHOP (Ro-CHOP) in the Treatment of Peripheral T-Cell Lymphomas
Brief Title: A Study of Escalating Doses of Romidepsin in Association With CHOP in the Treatment of Peripheral T-Cell Lymphomas
Acronym: Ro-CHOP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ro-CHOP
Record Dates: First submitted 2011-01-14; First posted 2011-01-20 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Romidepsin dose 10mg/m² (Experimental): Romidepsin dose 10mg/m²
  Interventions: Drug: Romidepsin and CHOP
- Romidepsin dose 12mg/m² (Experimental): Romidepsin dose 12mg/m²
  Interventions: Drug: Romidepsin and CHOP
- Romidepsin dose 14mg/m² (Experimental): Romidepsin dose 14mg/m²
  Interventions: Drug: Romidepsin and CHOP
- Romidepsin dose 8mg/m² (Experimental): Romidepsin dose 8mg/m²
  Interventions: Drug: Romidepsin and CHOP

INTERVENTIONS:
Drug: Romidepsin and CHOP — Romidepsin dose administered IV at day 1 and 8 or at day 1 without day 8 in combination with cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered every 3 weeks for 8 cycles in patients with T-cell lymphoma
  Arms: Romidepsin dose 10mg/m²
Drug: Romidepsin and CHOP — Romidepsin dose administered IV at day 1 and 8 or at day 1 without day 8 in combination with cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered every 3 weeks for 8 cycles in patients with T-cell lymphoma
  Arms: Romidepsin dose 12mg/m²
Drug: Romidepsin and CHOP — Romidepsin dose administered IV at day 1 and 8 or at day 1 without day 8 in combination with cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered every 3 weeks for 8 cycles in patients with T-cell lymphoma
  Arms: Romidepsin dose 14mg/m²
Drug: Romidepsin and CHOP — Romidepsin dose administered IV at day 1 and 8 or at day 1 without day 8 in combination with cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered every 3 weeks for 8 cycles in patients with T-cell lymphoma
  Arms: Romidepsin dose 8mg/m²

SUMMARY:
This study is an open label, multicenter study with two phases:

* A dose escalation phase of Romidepsin administered IV at day 1 and 8 or at day 1 without day 8 in combination with cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP)administered every 3 weeks for 8 cycles in patients with T-cell lymphoma.
* An expansion phase in order to assess the safety and the efficacy of the association of the recommended dose of Romidepsin associated with CHOP in a population of patients with T-cell lymphoma.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the feasibility of the combination and the recommended dose (RD) of Romidepsin when administered in association with CHOP in a population of patients with newly diagnosed Peripheral T-cell lymphoma (PTCL) as measured by the toxicities during treatment.

Secondary objectives:

* To assess the safety of the association Romidepsin and CHOP,
* To assess the efficacy of the association of Romidepsin and CHOP: response rate and complete response rate, progression-free survival, response duration and overall survival.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Patients with histologically confirmed Peripheral T-cell Lymphoma (PTCL), not previously treated ; all subtypes may be included except HTLV-1-related T-cell lymphoma, cutaneous T-cell lymphoma (mycosis fungoid and Sézary syndrome), and ALK+ PTCL,
   2. Ann Arbor stages II - IV
   3. Aged from 18 to 80 years,
   4. ECOG performance status 0, 1 or 2,
   5. Signed informed consent,
   6. Negative pregnancy test for females of childbearing potential (FCBP),
   7. FCBP using an effective method of birth control (i.e. hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide or abstinence) for the treatment period and for 1 month thereafter; Males using an effective method of birth control for the treatment period and 3 months thereafter,
   8. Life expectancy of ≥ 90 days (3 months)
2. Exclusion Criteria:

   1. Other types of lymphomas, e.g. B-cell lymphoma
   2. Ann Arbor stage I
   3. Previous treatment for PTCL with immunotherapy or chemotherapy except for short-term corticosteroids before inclusion
   4. Previous radiotherapy for PTCL except if localized to one lymph node area
   5. Central nervous system - meningeal involvement
   6. Contraindication to any drug contained in the chemotherapy regimen
   7. HIV infection, active hepatitis B or C
   8. Any serious active disease or co-morbid medical condition (according to investigator's decision)
   9. Any of the following laboratory abnormalities

      * Absolute neutrophil count (ANC) < 1,500 cells/mm3 (1.5 x 109/L),
      * Platelet count < 100,000/mm3 (100 x 109/L), or 75,000 if bone marrow is involved,
      * Serum SGOT/AST or SGPT/ALT ≥ 5.0 x upper limit of normal (ULN),
      * Serum total bilirubin > 2.0 mg/dL (34 µmol/L), except in case of hemolytic anemia,
      * Low K+ (inferior to low normal level) and low Mg+ (inferior to low normal level)levels, except if corrected before beginning the chemotherapy,
   10. Use of oral contraceptive and contraceptive patches,
   11. Calculated creatinine clearance (Cockcroft-Gault formula) of < 50 mL /min,
   12. Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 3 years,
   13. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form,
   14. Left Ventricular Ejection Fraction < 45% (calculated by echocardiographic or scintigraphic methods),
   15. Patients with congenital long QT syndrome, history of significant cardiovascular disease and/or taking drugs leading to significant QT prolongation,
   16. Corrected QT interval > 480 msec (using the fridericia formula)
   17. Use of any standard or experimental anti-cancer drug therapy within 28 days of the initiation (Day 1) of study drug ,
   18. Pregnant or lactating females or women of childbearing potential not will-ing to use an adequate method of birth control for the duration of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | 42 days

SECONDARY OUTCOMES:
Complete Response Rate(CR) at the end of treatment | 30 days after the end of treatment
Progression-free survival (PFS) | from the date of inclusion to the date of first documentated disease progression, relapse or death from any cause
Duration of Response | from the date of first documentation of a response to the date of first documented evidence of progression/relapse or death from any cause
Safety of association Romidepsin-CHOP | from the date of informed consent signature to 90 days after the last drug administration
  Toxicities occured during the trial for all patient from the date of informed consent signature to 90 days after the last drug administration will be measured and reported for all grades toxicities according to CTCAE v4.
Overall Response at the end of treatment | 30 days after the end of treatment
Overall Survival (OS) | from the date of inclusion to the date of first documentated disease progression, relapse or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand COIFFIER, Professor, Principal Investigator
Locations (8):
- France (8):
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - Hôpital Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital St Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Dupuis J, Morschhauser F, Ghesquieres H, Tilly H, Casasnovas O, Thieblemont C, Ribrag V, Bossard C, Le Bras F, Bachy E, Hivert B, Nicolas-Virelizier E, Jardin F, Bastie JN, Amorim S, Lazarovici J, Martin A, Coiffier B. Combination of romidepsin with cyclophosphamide, doxorubicin, vincristine, and prednisone in previously untreated patients with peripheral T-cell lymphoma: a non-randomised, phase 1b/2 study. Lancet Haematol. 2015 Apr;2(4):e160-5. doi: 10.1016/S2352-3026(15)00023-X. Epub 2015 Mar 17. PMID 26687958